CLINICAL TRIAL: NCT06685458
Title: Combined With Clinical and Imaging Features, the Prediction Model of Benign and Malignant Solid Pulmonary Nodules Was Constructed
Brief Title: Constructing a Predictive Model for Differentiating Between Benign and Malignant Solid Pulmonary Nodules Based on Clinical and Imaging Features.
Status: Not yet recruiting | Type: Observational
Sponsor: The Third Affiliated Hospital of Kunming Medical College. (Other)
Responsible Party: Principal Investigator, Yantao Yang, Physician, The Third Affiliated Hospital of Kunming Medical College.
Other Study IDs: KYLX2024-271
Record Dates: First submitted 2024-11-10; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer; Solid Pulmonary Nodules; Pulmonary Nodules
Keywords: Lung Cancer Screening; Nodule Malignancy Prediction; Preoperative Imaging Analysis
MeSH Terms: conditions — Lung Neoplasms; Multiple Pulmonary Nodules

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Benign Nodule Group: Participants with benign solid pulmonary nodules.
  Interventions: Other: Preoperative Clinical and Imaging Feature Evaluation for Predictive Modeling
- Malignant Nodule Group: Participants with malignant solid pulmonary nodules.
  Interventions: Other: Preoperative Clinical and Imaging Feature Evaluation for Predictive Modeling

INTERVENTIONS:
Other: Preoperative Clinical and Imaging Feature Evaluation for Predictive Modeling — This study involves preoperative evaluation of clinical and imaging features for constructing a predictive model to differentiate benign and malignant solid pulmonary nodules. Surgical resection is performed to obtain pathological confirmation as the reference standard.

SUMMARY:
Study Objective:

To comprehensively analyze the preoperative clinical and imaging characteristics of solid pulmonary nodules, investigate the risk factors associated with malignant solid pulmonary nodules, and provide a reference for preoperative treatment decisions.

Significance of the Study:

According to the 2020 Global Cancer Report, lung cancer remains the leading cause of cancer-related deaths worldwide. While the majority of patients with stage I lung cancer achieve long-term survival, survival rates for advanced-stage patients are extremely low. Early screening, diagnosis, and treatment of lung cancer are crucial.

With the widespread implementation of early lung cancer screening, a growing number of pulmonary nodules are being detected, among which solid pulmonary nodules constitute a significant proportion. Unlike ground-glass nodules, accurately distinguishing between benign and malignant solid nodules is critical for determining appropriate treatment strategies. For benign solid nodules, follow-up observation is the preferred approach, whereas early surgical intervention is essential for malignant solid nodules.

Although previous studies have explored the correlation between clinical and imaging characteristics, they have not conducted systematic analyses, and most have been based on small sample sizes. Therefore, this study aims to conduct a comprehensive analysis of preoperative clinical and imaging characteristics, build a predictive model to differentiate between benign and malignant solid pulmonary nodules, and provide a reliable reference for selecting treatment strategies.

DETAILED DESCRIPTION:
Our study evaluate patients with SPN from the Third Affiliated Hospital of Kunming Medical University. The patient selection followed specific inclusion and exclusion criteria. Inclusion criteria included: (1) All subjects provided CT imaging obtained from the Third Affiliated Hospital of Kunming Medical University within 2-week period prior to surgery; (2) Complete clinicopathological data of solid nodules were obtained; (3) Surgical intervention for one or more SPN; (4) No prior anti-tumor treatments like radiotherapy or chemotherapy; (5) Age 18 years or older. Exclusion criteria involved: (1) Patients with incomplete imaging data or medical records; (2) Lung infections that could affect image analysis; (3) Significant respiratory movement artifacts in images impairing imaging analysis; (4) Inconsistent locations of SPN in postoperative pathology reports and preoperative CT images.

ELIGIBILITY:
Inclusion Criteria:

* (1) All subjects provided CT imaging obtained from the Third Affiliated Hospital of Kunming Medical University within 2-week period prior to surgery; (2) Complete clinicopathological data of solid nodules were obtained; (3) Surgical intervention for one or more SPN; (4) No prior anti-tumor treatments like radiotherapy or chemotherapy; (5) Age 18 years or older.

Exclusion Criteria:

* (1) Patients with incomplete imaging data or medical records; (2) Lung infections that could affect image analysis; (3) Significant respiratory movement artifacts in images impairing imaging analysis; (4) Inconsistent locations of SPN in postoperative pathology reports and preoperative CT images.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients aged 18 years and older with radiologically diagnosed solid pulmonary nodules. These patients are undergoing preoperative clinical and imaging evaluations and subsequent surgical resection to confirm the benign or malignant nature of the nodules
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of predictive model | Within 2 years after surgical resection and pathological confirmation
  The primary outcome is the area under the receiver operating characteristic curve (AUC) of the predictive model in distinguishing benign from malignant solid pulmonary nodules, based on preoperative clinical and imaging features.

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due sharing data is not included in our research institution review board.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Goldstraw P, Chansky K, Crowley J, Rami-Porta R, Asamura H, Eberhardt WE, Nicholson AG, Groome P, Mitchell A, Bolejack V; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee, Advisory Boards, and Participating Institutions; International Association for the Study of Lung Cancer Staging and Prognostic Factors Committee Advisory Boards and Participating Institutions. The IASLC Lung Cancer Staging Project: Proposals for Revision of the TNM Stage Groupings in the Forthcoming (Eighth) Edition of the TNM Classification for Lung Cancer. J Thorac Oncol. 2016 Jan;11(1):39-51. doi: 10.1016/j.jtho.2015.09.009. PMID 26762738
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Choo E. Testing: High-Resolution Chest Computed Tomography Scan. Springer New York. 2014.
- [Background] Yip R, Li K, Liu L, Xu D, Tam K, Yankelevitz DF, Taioli E, Becker B, Henschke CI. Controversies on lung cancers manifesting as part-solid nodules. Eur Radiol. 2018 Feb;28(2):747-759. doi: 10.1007/s00330-017-4975-9. Epub 2017 Aug 23. PMID 28835992
- [Background] Winer-Muram HT. The solitary pulmonary nodule. Radiology. 2006 Apr;239(1):34-49. doi: 10.1148/radiol.2391050343. PMID 16567482
- [Background] McWilliams A, Tammemagi MC, Mayo JR, Roberts H, Liu G, Soghrati K, Yasufuku K, Martel S, Laberge F, Gingras M, Atkar-Khattra S, Berg CD, Evans K, Finley R, Yee J, English J, Nasute P, Goffin J, Puksa S, Stewart L, Tsai S, Johnston MR, Manos D, Nicholas G, Goss GD, Seely JM, Amjadi K, Tremblay A, Burrowes P, MacEachern P, Bhatia R, Tsao MS, Lam S. Probability of cancer in pulmonary nodules detected on first screening CT. N Engl J Med. 2013 Sep 5;369(10):910-9. doi: 10.1056/NEJMoa1214726. PMID 24004118
- [Background] Sim YT, Goh YG, Dempsey MF, Han S, Poon FW. PET-CT evaluation of solitary pulmonary nodules: correlation with maximum standardized uptake value and pathology. Lung. 2013 Dec;191(6):625-32. doi: 10.1007/s00408-013-9500-6. Epub 2013 Sep 8. PMID 24013495
- [Background] Chu ZG, Zhang Y, Li WJ, Li Q, Zheng YN, Lv FJ. Primary solid lung cancerous nodules with different sizes: computed tomography features and their variations. BMC Cancer. 2019 Nov 7;19(1):1060. doi: 10.1186/s12885-019-6274-0. PMID 31699047
- [Background] Ye T, Deng L, Wang S, Xiang J, Zhang Y, Hu H, Sun Y, Li Y, Shen L, Xie L, Gu W, Zhao Y, Fu F, Peng W, Chen H. Lung Adenocarcinomas Manifesting as Radiological Part-Solid Nodules Define a Special Clinical Subtype. J Thorac Oncol. 2019 Apr;14(4):617-627. doi: 10.1016/j.jtho.2018.12.030. Epub 2019 Jan 17. PMID 30659988
- [Background] Sun K, You A, Wang B, Song N, Wan Z, Wu F, Zhao W, Zhou F, Li W. Clinical T1aN0M0 lung cancer: differences in clinicopathological patterns and oncological outcomes based on the findings on high-resolution computed tomography. Eur Radiol. 2021 Oct;31(10):7353-7362. doi: 10.1007/s00330-021-07865-2. Epub 2021 Apr 15. PMID 33860370
- [Background] Zhao WJ. Preliminary study on CT radiomics to differentiate tuberculosis, adenocarcinoma, and non-tuberculous infectious lesions manifesting as solid pulmonary nodules or masses. 2024.
- [Background] Li M, Han R, Song W, Wang X, Guo F, Su D, Yu T, Wang Y. [Three Dimensional Volumetric Analysis of Solid Pulmonary Nodules on Chest CT: Cancer Risk Assessment]. Zhongguo Fei Ai Za Zhi. 2016 May 20;19(5):279-85. doi: 10.3779/j.issn.1009-3419.2016.05.05. Chinese. PMID 27215456
- [Background] Ma X. Development and validation of a combined model based on imaging features and circulating tumor cells for differentiating benign and malignant solid pulmonary nodules. 2024.
- [Background] Zhu LL. Analysis of malignant risk factors and imaging and tumor marker expression characteristics in patients with solitary pulmonary nodules. 2022.